CLINICAL TRIAL: NCT01514266
Title: Effect of Curcumin on Lung Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Amir Sharafkhaneh, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-17419
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: proven diagnosis; COPD; sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin+bioprine (Experimental): The study involves active arm of Curcumin+Bioprine
  Interventions: Drug: Curcumin+Bioprine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin+Bioprine — The intervention arm is Curcumin+Bioprine at escalating doses of 1 gram of Curcumin and 5 mg of Bioprine bid for one month, then 1.5 grams of Curcumin and 5 mg of bioprine bid for one month, and finally 2 grams of curcumin with 5 mg of bioprine bid for additional one month.
  Arms: Curcumin+bioprine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) and lung cancer are leading causes of death and health care use. Diffuse airways inflammation is seen in COPD and is thought to be the reason for deterioration of lung function in COPD. Currently there is no medication available that can modify or reduce this inflammation. Furthermore, from literature review it has been shown that chronic inflammation can result in cancerous changes.

Curcumin is a food additive used for centuries. Several studies showed that curcumin suppress the different inflammatory pathways. Specially, the TNF-alpha and the NF kappa-b are down regulated by this substance. This study was designed to evaluate effect of combination of curcumin+Bioprine on sputum cytology in patients with COPD. This is double-blind randomized pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 45 with moderate COPD: FEV1/FVC ratio less than 70 percent; post bronchodilator FEV1 less than 50 percent
* 20 pack year cigarette smoking
* Stable clinical course (symptoms/ medications) for 8 weeks
* Fixed address/Not planning to leave
* Being able to perform spirometry
* Able to understand and consent

Exclusion Criteria:

* Other chronic respiratory diseases such as asthma, interstitial fibrosis, sarcoidosis
* Heart failure NYH III & IV; symptomatic liver or renal failure
* Dementia or other neurocognitive deficit preventing completion of symptom diary
* Use of inhaled or systemic corticosteroids within 8 weeks of enrollment in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in sputum dysplasia | 3 months
  We evaluated presence of moderate or worse dysplasia at baseline and each subsequent visits. The primary endpoint of this study is change in sputum cytological abnormality (moderate or worse dysplasia). The change will be comparison of 3-month follow up compared to baseline.

SECONDARY OUTCOMES:
Number of subjects with adverse events in each arm of the study. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center, Houston, Texas, United States